CLINICAL TRIAL: NCT00560352
Title: A Phase I Study of Dasatinib With Bortezomib (Velcade®) and Dexamethasone in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: Safety Study of Dasatinib With Bortezomib (Velcade®) and Dexamethasone for Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA180-181
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Results first posted 2012-07-09 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2012-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dasatinib; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dasatinib + Bortezomib + Dexamethasone (Experimental): Phase I dose escalation study
  Interventions: Drug: Dasatinib; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Dasatinib — Tablets; oral; approximately 2 years on study, depending on response; 50 mg once daily (QD), 100 mg QD, 140 mg QD
  Other Names: Sprycel; BMS-354825
Drug: Bortezomib — Powder; intravenous; approximately 2 years on study, depending on response; 1.0 mg/m^2 QD, 1.3 mg/m^2 QD
  Other Names: Velcade®
Drug: Dexamethasone — Tablets; oral; approximately 2 years on study, depending on response; 20 mg QD

SUMMARY:
The purpose of this study is to determine the safety and tolerability of dasatinib with bortezomib in the treatment of relapsed or refractory multiple myeloma.

ELIGIBILITY:
Key Inclusion Criteria:

* Confirmed diagnosis of multiple myeloma with measurable disease
* Evidence of relapsed or refractory disease and at least 2 prior therapies for multiple myeloma
* Eastern Cooperative Oncology Group Performance Status of 0 - 2
* Last treatment for multiple myeloma not within 21 days prior to study treatment initiation
* Bone marrow transplant not within 3 months prior to study treatment initiation
* Required baseline hematology and chemistry parameters.

Key Exclusion Criteria:

* Clinically significant cardiac disease (New York Heart Association Class III or IV)
* Abnormal QT interval corrected for heart rate using Fridericia's formula prolonged (>450 msec) after electrolytes have been corrected on baseline electrocardiogram
* Malabsorption syndrome or uncontrolled gastrointestinal toxicities
* Dementia, chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation
* Clinically significant pleural effusion in the previous 12 months or current ascites
* Clinically significant coagulation or platelet function disorder
* Intolerance to dasatinib and/or bortezomib
* Acute diffuse infiltrative pulmonary disease
* Prior or concurrent malignancy, except for adequately treated basal cell or squamous cell skin cancer, adequately treated Stage I or II cancer currently in complete remission, cervical carcinoma in situ, or any other cancer from which the participant has been disease-free for 3 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (7):
- United States (2):
  - Orlando Health, Inc. M.D. Anderson Cancer Center Orlando, Orlando, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
- France (2):
  - Local Institution, Nantes, Cedex 1
  - Local Institution, Lille
- Italy (2):
  - Local Institution, Bari
  - Local Institution, Bologna
- Local Institution, Salamanca, Spain

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 16 participants were enrolled, and 14 participants received treatment. The study was terminated due to an unexpectedly low recruitment rate, and no participants were enrolled in a planned dose-expansion phase.
Groups:
- Dasatinib, 50 mg BID: Dasatinib, 50 mg administered twice daily (BID), with 1.0 mg/m^2 of bortezomib in 21-day cycles. Dexamethasone, fixed at 20 mg once daily (QD), was administered the day of and 1 day after each bortezomib dosing. In a 21-day cycle, bortezomib was administered by intravenous (IV) bolus twice weekly, on Days 1, 4, 8, and 11, followed by a 10-day (Days 12 to 21) rest period. In a 21-day cycle, dasatinib was taken orally every day, BID. In a 21-day cycle, dexamethasone was taken orally on Days 1, 2, 4, 5, 8, 9, 11, and 12, at the same time as dasatinib. On the days when bortezomib and dasatinib were administered together, the morning dose of dasatinib was to be followed 1-2 hours by the dose of bortezomib.
- Dasatinib, 100 mg QD: Dasatinib, 100 mg, given QD with 1.3 mg/m^2 of bortezomib in 21-day cycles. Dexamethasone, fixed at 20 mg QD, was administered the day of and 1 day after each bortezomib dosing. In a 21-day cycle, bortezomib was administered by IV bolus twice weekly, on Days 1, 4, 8, and 11, followed by a 10-day (Days 12 to 21) rest period. In a 21-day cycle, dasatinib was taken orally every day, QD in the morning. In a 21-day cycle, dexamethasone was taken orally on Days 1, 2, 4, 5, 8, 9, 11, and 12, at the same time as dasatinib. On the days when bortezomib and dasatinib were administered together, the morning dose of dasatinib was to be followed 1-2 hours by the dose of bortezomib.
- Dasatinib, 140 mg QD: Dasatinib, 140 mg, administered QD with 1.3 mg/m^2 of bortezomib in 21-day cycles. Dexamethasone, fixed at 20 mg QD, was administered the day of and 1 day after each bortezomib dosing.In a 21-day cycle, bortezomib was administered by IV bolus twice weekly, on Days 1, 4, 8, and 11, followed by a 10-day (Days 12 to 21) rest period. In a 21-day cycle, dasatinib was taken orally every day, QD in the morning. In a 21-day cycle, dexamethasone was taken orally on Days 1, 2, 4, 5, 8, 9, 11, and 12, at the same time as dasatinib. On the days when bortezomib and dasatinib were administered together, the morning dose of dasatinib was to be followed 1-2 hours by the dose of bortezomib.
Period: Overall Study
Arm/Group | Dasatinib, 50 mg BID | Dasatinib, 100 mg QD | Dasatinib, 140 mg QD
Started | 7 | 3 | 4
Completed | 0 | 0 | 0
Not Completed | 7 | 3 | 4
Not completed — Adverse event unrelated to study drug | 2 | 1 | 1
Not completed — Study drug toxicity | 3 | 0 | 1
Not completed — Disease progression | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Maximum clinical benefit | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dasatinib, 50 mg BID | Dasatinib, 100 mg QD | Dasatinib, 140 mg QD | Total
Number analyzed (Participants) | 7 | 3 | 4 | 14
Age, Continuous [Mean (Full Range); unit: Years] | 72 [64.0 to 74.0] | 74 [57.0 to 75.0] | 59.5 [53.0 to 75.0] | 71 [53.0 to 75.0]
Age, Customized [Number; unit: Participants]
  46 to 65 years | 1 | 1 | 3 | 5
  66 to 75 years | 6 | 2 | 1 | 9
  Older than 75 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 6
  Male | 5 | 2 | 1 | 8
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 6 | 3 | 4 | 13
  Black or African American | 0 | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Other | 1 | 0 | 0 | 1
  Not reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) and Recommended MTD of Dasatinib in Combination With Bortezomib and Dexamethasone
Description: MTD is defined as the dose level combination below the dose level that produces a dose-limiting toxicity in at least 2 out of 6 or fewer participants in that cohort. If MTD is not reached, the recommended MTD is the maximum dose that the participants received.
Time Frame: Days 1 to 21
Population: All participants who received at least 1 dose of dasatinib and/or bortezomib and/or dexamethasone
Measure: Number; unit: mg QD
Groups:
- All Treated: Dasatinib taken orally every day, once daily (QD) or twice daily (BID), depending on the assigned cohort dose level, in 21-day cycles. In a 21-day cycle, bortezomib was also administered by intravenous (IV) bolus twice weekly, on Days 1, 4, 8, and 11, followed by a 10-day (Days 12 to 21) rest period. In a 21-day cycle, dexamethasone was taken orally on Days 1, 2, 4, 5, 8, 9, 11, and 12, at the same time as dasatinib. On the days when bortezomib and dasatinib were administered together, the morning dose of dasatinib was followed 1-2 hours later by the dose of bortezomib. In the dose-escalation phase (Part 1), participants were enrolled sequentially in groups of 3 and individually assessed for safety and dose-limiting toxicity.
Arm/Group | All Treated
Number analyzed (Participants) | 14
mg QD
  MTD dasatinib | NA — The MTD was not reached at the highest dose level defined by protocol for this study.
  Recommended MTD dasatinib | 140

2. Secondary Outcome: Best Overall Tumor Response Rate (RR) As Assessed Using International Uniform Response Criteria for Multiple Myeloma and Criteria of the European Bone Marrow Transplant Registry
Description: S=serum; U=urine; MP=M-protein; ST=soft tissue, PC=plasmacytomas; IF=immunofixation; BL=baseline. RR calculated on best response any time. CR=MP undetectable by IF, ≤5% plasma cells in bone marrow, and no ST PC. VGPR=MP detectable by IF, or ≥90% drop in S MP and U MP<100 mg/24h. PR= ≥50% drop in S MP and ≥90% drop in U MP or U protein <200 mg/24h, ≥50% drop in BL ST PC size. MR= ≥25% to <50% drop in S MP and ≥50% to <90% drop in U MP and ≥25% to <50% drop in BL ST PC. SD=Not CR, VGPR, PR, or MR. PD= ≥25% rise in S or U M-component; new/increased size of bone lesions, ST PC, or hypercalcemia.
Time Frame: Day 1 until last tumor assessment (maximum reached: 9 months)
Population: All response-evaluable participants who received at least 1 dose of dasatinib and/or bortezomib and/or dexamethasone
Measure: Number; unit: Percentage of participants
Arm/Group | Dasatinib, 50 mg BID | Dasatinib, 100 mg QD | Dasatinib, 140 mg QD
Number analyzed (Participants) | 7 | 3 | 4
Percentage of participants
  Complete response (CR) | 0 | 0 | 0
  Very good partial response (VGPR) | 0 | 0 | 0
  Partial response (PR) | 14.3 | 0 | 0
  Minimal response (MR) | 0 | 0 | 25
  Stable disease (SD) | 57.1 | 0 | 0
  Progressive disease (PD) | 14.3 | 33.3 | 0
  Unable to determine | 0 | 33.3 | 25
  Not reported | 14.3 | 33.3 | 50

3. Secondary Outcome: Duration of Response
Description: Duration of response calculated for those with best response=CR (M-protein [MP] undetectable by immunofixation [IF], ≤5% plasma cells in bone marrow, no soft tissue plasmacytomas); VGPR (MP detectable by IF, or ≥90% drop in serum [S] MP and urine [U] MP<100 mg/24h); PR(≥50% drop in S MP and ≥90% drop in U MP or U protein <200 mg/24h, ≥50% drop in BL ST PC size); or MR (≥25% to <50% drop in S MP and ≥50% to <90% drop in U MP and ≥25% to <50% drop in BL ST PC). Duration of response calculated from day criteria for CR, VGPR, PR, and MR were met until progression or death, whichever came first.
Time Frame: First occurrence of response to disease progression or death, whichever occurred first (maximum reached: 12.2 months)
Population: All response-evaluable participants who achieved a response.
Measure: Number; unit: Months
Groups:
- Dasatinib, 50 mg BID: Dasatinib, 50 mg administered BID, with 1.0 mg/m^2 of bortezomib in 21-day cycles. Dexamethasone, fixed at 20 mg QD, was administered the day of and 1 day after each bortezomib dosing. In a 21-day cycle, bortezomib was administered by IV bolus twice weekly, on Days 1, 4, 8, and 11, followed by a 10-day (Days 12 to 21) rest period. In a 21-day cycle, dasatinib was taken orally every day, BID. In a 21-day cycle, dexamethasone was taken orally on Days 1, 2, 4, 5, 8, 9, 11, and 12, at the same time as dasatinib. On the days when bortezomib and dasatinib were administered together, the morning dose of dasatinib was to be followed 1-2 hours by the dose of bortezomib.
Arm/Group | Dasatinib, 50 mg BID | Dasatinib, 100 mg QD | Dasatinib, 140 mg QD
Number analyzed (Participants) | 1 | 0 | 1
Months
  Partial response (PR) | 5.4 |  | 0
  Minimal response (MR) | NA — There were 0 participants who received 50 mg BID of dasatanib who had a minimal response. |  | 12.2

4. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from start of treatment until progression or death, whichever occurred first. Participants were to be followed-up for 12 months following the last dose of dasatinib for progression and survival. PFS was analyzed for the all-treated population.
Time Frame: Day 1 to disease progression or death, whichever came first (maximum reached: 14 months)
Population: All participants who received at least 1 dose of dasatinib and/or bortezomib and/or dexamethasone
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- All Treated: Dasatinib taken orally every day, QD or BID, depending on the assigned cohort dose level, in 21-day cycles. In a 21-day cycle, bortezomib was also administered by IV bolus twice weekly, on Days 1, 4, 8, and 11, followed by a 10-day (Days 12 to 21) rest period. In a 21-day cycle, dexamethasone was taken orally on Days 1, 2, 4, 5, 8, 9, 11, and 12, at the same time as dasatinib. On the days when bortezomib and dasatinib were administered together, the morning dose of dasatinib was followed 1-2 hours later by the dose of bortezomib. In the dose-escalation phase (Part 1), participants were enrolled sequentially in groups of 3 and individually assessed for safety and dose-limiting toxicity.
Arm/Group | All Treated
Number analyzed (Participants) | 14
Months | 6.3 [2.4 to 14.0]

5. Secondary Outcome: Number of Participants With Death As Outcome, Serious Adverse Events (SAEs), Drug-related SAEs, Drug-related Adverse Events (AEs) Leading to Discontinuation, AEs Leading to Discontinuation, AEs, and Drug-related AEs by Grade
Description: An AE is any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that does not necessarily have a causal relationship with treatment. An SAE is any unfavorable medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency or abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Drug-related=possibly, probably, or certainly related to or of unknown relationship to study treatment. Grade 3=severe; Grade 4=life-threatening.
Time Frame: Continuously from Day 1 until last day of study medication + 30 days (maximum reached: 10 months)
Population: All participants who received at least 1 dose of dasatinib and/or bortezomib and/or dexamethasone.
Measure: Number; unit: Participants
Groups:
- Dasatinib, 50 mg BID: Dasatinib, 50 mg administered BID, with 1.0 mg/m^2 of bortezomib in 21-day cycles. Dexamethasone, fixed at 20 mg QD, was administered the day of and 1 day after each bortezomib dosing. In a 21-day cycle, bortezomib was administered by intravenous (IV) bolus twice weekly, on Days 1, 4, 8, and 11, followed by a 10-day (Days 12 to 21) rest period. In a 21-day cycle, dasatinib was taken orally every day, BID. In a 21-day cycle, dexamethasone was taken orally on Days 1, 2, 4, 5, 8, 9, 11, and 12, at the same time as dasatinib. On the days when bortezomib and dasatinib were administered together, the morning dose of dasatinib was to be followed 1-2 hours by the dose of bortezomib.
Arm/Group | Dasatinib, 50 mg BID | Dasatinib, 100 mg QD | Dasatinib, 140 mg QD
Number analyzed (Participants) | 7 | 3 | 4
Participants
  Death | 3 | 2 | 2
  SAEs | 6 | 2 | 1
  Drug-related SAEs | 2 | 0 | 0
  Drug-related AEs leading to discontinuation | 3 | 0 | 1
  AEs leading to discontinuation | 5 | 1 | 2
  AEs | 7 | 3 | 4
  AEs, Grades 3 and 4 | 3 | 3 | 4
  Drug-related AEs | 6 | 2 | 4
  Drug-related AEs, Grades 3 and 4 | 4 | 2 | 4

6. Primary Outcome: MTD and Recommended MTD of Bortezomib in Combination With Dasatinib and Dexamethasone
Description: MTD is defined as the dose level combination below the dose level that produces a dose-limiting toxicity in at least 2 out of 6 or fewer participants in that cohort. If MTD is not reached, the recommended dose is the maximum dose that the participants received.
Time Frame: Days 1 to 21
Population: All participants who received at least 1 dose of dasatinib and/or bortezomib and/or dexamethasone
Measure: Number; unit: mg/m^2
Arm/Group | All Treated
Number analyzed (Participants) | 14
mg/m^2
  MTD of bortezomib | NA — The MTD was not reached at the highest dose level defined by protocol for this study.
  Recommended MTD of bortezomib | 1.3

ADVERSE EVENTS:
Time Frame: Continuously from Day 1 until last day of study medication + 30 days (maximum reached: 10 months)
Arm/Group | Dasatinib, 100 mg QD | Dasatinib, 140 mg QD | Dasatinib, 50 mg BID
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/4 | 6/7
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib, 100 mg QD (N=3) | Dasatinib, 140 mg QD (N=4) | Dasatinib, 50 mg BID (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib, 100 mg QD (N=3) | Dasatinib, 140 mg QD (N=4) | Dasatinib, 50 mg BID (N=7)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 4
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 2
Irritability (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 3
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Gastrointestinal candidiasis (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1
Nocturia (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Urine flow decreased (Renal and urinary disorders) | 1 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated due to an unexpectedly low recruitment rate, and no participants were enrolled in a planned dose-expansion phase.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.